CLINICAL TRIAL: NCT04133181
Title: Clinical and Radiographic Success of Guided Versus Conventional Periapical Endodontic Surgery: A Randomized Controlled Trial
Brief Title: Guided Versus Conventional Periapical Endodontic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, ahmed meneisy, Doctor Degree candidate, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Endosurgery
Record Dates: First submitted 2019-10-17; First posted 2019-10-21 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Endodontic Disease; Endodontic Re-treatment Failure
Keywords: Endodontic surgery; Guided surgery; 3D guide
MeSH Terms: conditions — Dental Pulp Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Guided endodontic surgery (Experimental): Use of a 3D surgical guide in endodontic surgery
  Interventions: Device: 3D guide
- Conventional endodontic surgery (Placebo Comparator): Use of a mock guide in endodontic surgery
  Interventions: Device: Mock guide

INTERVENTIONS:
Device: 3D guide — Use of a 3D guide in endodontic surgery
  Arms: Guided endodontic surgery
Device: Mock guide — Use of a mock guide in endodontic surgery
  Arms: Conventional endodontic surgery

SUMMARY:
This study is to compare the clinical and radiographic outcomes after guided periapical endodontic surgery versus conventional endodontic surgery.

DETAILED DESCRIPTION:
The aim of this study is to compare the clinical and radiographic outcomes after guided periapical endodontic surgery versus conventional endodontic surgery. Patients having mandibular posterior teeth indicated for endodontic surgery will be selected. Full medical and dental history will be obtained from all patients. Patients will be randomly assigned to either guided endodontic surgery or conventional endodontic surgery. Surgical procedures will be done under magnification. Root-end cavities will be filled using MTA.Post surgical instrucions will be given to patients. Surgical time will be recorded. Clinical and radiographic success will be asses at 6 and 12 month.

ELIGIBILITY:
Inclusion Criteria:

1. Patients in good general health.
2. Patients with age ranging between 18-50 years with no sex predilection.
3. Posterior teeth with an indication for endodontic surgery.
4. Patients' acceptance to participate in the study.

Exclusion Criteria:

1. Patients with allergy to materials or medications used in the trial.
2. Pregnant female patients.
3. Teeth with pathoses associated with vertical root fracture.
4. Severe periodontal bone loss detected with a periodontal probe (5 mm probing depth).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Clinical success | 1 year
  Clinical assessment using a scale by friedman et al 2005 (healed, healing and persisting disease) which healed mean absence of clinical signs and symptoms, persisting disease mean presence of clinical signs and symptoms
Radio graphic Success | 1 year
  Radiograhic assessment using a scale by friedman et al 2005 (healed, healing and persisting disease) which healed mean radiographic classification of complete healing or incomplete healing, persisting disease mean radiographic classification of unsatisfactory healing.

SECONDARY OUTCOMES:
Time of surgery | During surgery
  Recording the surgical time in minutes.

REFERENCES:
- [Background] Anderson J, Wealleans J, Ray J. Endodontic applications of 3D printing. Int Endod J. 2018 Sep;51(9):1005-1018. doi: 10.1111/iej.12917. Epub 2018 Mar 23. PMID 29486052
- [Background] Strbac GD, Schnappauf A, Giannis K, Moritz A, Ulm C. Guided Modern Endodontic Surgery: A Novel Approach for Guided Osteotomy and Root Resection. J Endod. 2017 Mar;43(3):496-501. doi: 10.1016/j.joen.2016.11.001. Epub 2017 Jan 28. PMID 28139285
- [Background] Ahn SY, Kim NH, Kim S, Karabucak B, Kim E. Computer-aided Design/Computer-aided Manufacturing-guided Endodontic Surgery: Guided Osteotomy and Apex Localization in a Mandibular Molar with a Thick Buccal Bone Plate. J Endod. 2018 Apr;44(4):665-670. doi: 10.1016/j.joen.2017.12.009. Epub 2018 Jan 19. PMID 29358006